CLINICAL TRIAL: NCT00877604
Title: A Randomized, Double-blind Multicenter Pilot Study vs. Placebo for the Evaluation of Efficacy and Tolerability of Tauroursodeoxycholic Acid Administered by Oral Route as Add on Treatment in Patients Affected by Amyotrophic Lateral Sclerosis
Brief Title: Efficacy and Tolerability of Tauroursodeoxycholic Acid in Amyotrophic Lateral Sclerosis
Acronym: TUDCA-ALS
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Fondazione I.R.C.C.S. Istituto Neurologico Carlo Besta (Other)
Collaborators: University of Palermo (Other); Federico II University (Other)
Responsible Party: Principal Investigator, Alberto Albanese, Professor, Fondazione I.R.C.C.S. Istituto Neurologico Carlo Besta
Allocation: Randomized | Model: Single Group | Masking: Quadruple | Purpose: Treatment
Other Study IDs: TUDCA200701; EudraCT No.: 2007-001592-10
Record Dates: First submitted 2009-04-07; First posted 2009-04-08 (Estimated); Results first posted 2014-11-26 (Estimated); Last update posted 2014-11-26 (Estimated); Status verified 2014-11

CONDITIONS: Amyotrophic Lateral Sclerosis
Keywords: ALS; Therapy; Tauroursodeoxycholic acid; TUDCA; antioxidant; antiapoptotic drug; neuroprotective drug
MeSH Terms: conditions — Amyotrophic Lateral Sclerosis | interventions — ursodoxicoltaurine; Ursodeoxycholic Acid; Drugs, Generic; WW Domain-Containing Oxidoreductase

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- TUDCA (Experimental): tauroursodeoxycholic acid di-hydrate
  Interventions: Drug: tauroursodeoxycholic acid (TUDCA)
- placebo (Placebo Comparator): excipient lactose
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: tauroursodeoxycholic acid (TUDCA) — Oral route at the dose of 1 g b.i.d. (2 g daily) for 1 year
  Other Names: Ursodiol; Actigall; Generic
  Arms: TUDCA
Drug: Placebo — identical placebo by oral route at the same dosing schedule
  Other Names: Oral route at the dose of 1 g b.i.d. (2 g daily) for 1 year
  Arms: placebo

SUMMARY:
The preclinical rationale for tauroursodeoxycholic acid (TUDCA) use in treating patients with amyotrophic lateral sclerosis (ALS) stems from the demonstration of antioxidant, antiapoptotic and neuroprotective properties of TUDCA in the central nervous system (CNS), both in vitro and in vivo models.

This protocol is meant for assessing if the addition of TUDCA to the conventional therapy can improve the therapeutic outcome in patients affected by ALS.

Safety will be assessed for all subjects, for the entire duration of the study. 30 patients affected by ALS with site of onset in the limbs will be recruited.

All enrolled subjects will continue receiving riluzole at the same regimen as before entering the trial. Based on an appropriate random code, subjects will be divided into two groups of equal size treated, after a lead-in period of 3 months, by oral route with TUDCA at the dose 2 g daily for 1 year or with identical placebo by oral route at the same dosing schedule, under double-blind conditions.

Every concomitant and/or supportive therapy will be admitted.

Evaluation criteria:

Efficacy. The proportion of responder patients in the two treatment groups was the primary outcome measure of the study. Responder patients were defined as those subjects showing an improvement of at least 15% in the ALSFRS-R (2) slope during the treatment period as compared to the lead-in period. This threshold was chosen based according to the consensus conference on designing and implementing clinical trials in ALS (3).

Other parameters will include ALSFRS-R at study end, FVC%, the SF-36 quality of life rating scale, time to tracheotomy from starting of study medication dosing (if appropriate), survival Time from starting of study medication dosing (if appropriate), Medical Research Council scores for right and left muscle groups.

Safety. Incidence, severity and type of adverse events; changes in clinical laboratory findings.

DETAILED DESCRIPTION:
Amyotrophic lateral sclerosis (ALS), or motor neuron disease (MND), is a rapidly progressive, fatal neurodegenerative condition characterized by loss of upper and lower motor neurons in the brain and spinal cord. The terms ALS and MND are often used inter-changeably to cover the different clinical syndromes, which include upper and lower motor neuron disorder, progressive bulbar palsy, and pseudo-polyneuritic form.

Degeneration of lower motor neurons (LMN) in the anterior horns of spinal cord and brainstem leads to progressive muscular atrophy and eventually to death within a few years due to respiratory insufficiency. During the course of the disease, the involvement of tongue and pharynx muscles causes swallowing impairment with marked drooling, need of parenteral or enteral feeding, and finally gastrostomy. Denervation of laryngeal muscles causes loss of speech. Cramps and fasciculation typically occur from the early phases of the disease. Degeneration of upper motor neurons (UMN) in the brain cortex causes pyramidal tract dysfunctions including clonus, Babinski sign, hypertonia, and loss of dexterity that further limit patients' daily activities.

The incidence of ALS varies from 0.2 to 2.5 cases per 100,000 per year, although estimates vary between countries, likely reflecting a combination of availability of medical services, diagnostic accuracy, and demo-graphic characteristics of the area. Increasing life expectancy and improvements in standards of treatment and care will also result in an increased incidence of ALS. Globally, the overall rate is approximately 2 per 100,000. Its prevalence is approximately of 7 per 100,000. In Italy, the reported incidence of ALS is 2.2 cases/100,000/year.

There is currently no cure for ALS. Despite initial positive results in preclinical and early clinical studies, large-scale clinical trials with all agents except riluzole failed to demonstrate a clinically meaningful therapeutic effect in patients with ALS. Riluzole at the dose of 100 mg/day showed a significant difference on survival (6.4%; gain of 3 months) and slowed deterioration in muscle strength.

Primary involvement of apoptotic mechanisms has important implications in selecting drug candidates for therapy in ALS. Recent preclinical studies have demonstrated that TUCA is endowed with antioxidant, antiapoptotic and neuroprotective activities. In particular, TUDCA can cross the blood-brain-barrier and has been shown to exert a significant therapeutic effect in a model of HD mice.

Tauroursodeoxycholic acid (TUDCA) is a hydrophilic bile acid that is normally produced endogenously in humans at very low levels. TUDCA is synthesized in the liver by conjugation of taurine to ursodeoxycholic acid (UDCA), which is commonly used as a bile acid replacement therapy for the treatment of certain cholestatic syndromes.

The main pharmacological activity of TUDCA consists in its ability in increasing the cholesterol solubilising activity of bile, thus transforming "lithogenic" bile in "non-lithogenic" or "litholytic" bile.

TUDCA inhibits mitochondrial-associated apoptosis via many pathways: 1) it inhibits the mitochondrial permeability transition (MPT) and cytochrome C release, 2) it inhibits mitochondrial membrane depolarization, and 3) it antagonizes Bax translocation from the mitochondria and caspase activation in hepatocytes and brain. TUDCA may also ease oxidative stress.Study relevant TUDCA pharmacology consists in its antioxidant, antiapoptotic and neuroprotective activities evidenced in preclinical studies.

Recent reports have shown that hydrophilic bile acids, such as UDCA and TUDCA, can prevent hepatic cytotoxicity through several mechanisms. For example, TUDCA prevents the production of reactive oxygen species and thus acts as an antioxidant. Additionally, TUDCA mitigates mitochondrial insufficiency and toxicity, and prevents apoptosis, in part, by inhibiting Bax translocation from cytosol to the mitochondria. In hepatocytes, this inhibition results in reduced mitochondrial membrane perturbation, release of cytochrome c, and activation of downstream caspases. TUDCA reduced cytotoxicity in neurons through similar mechanisms, as well as mitochondrial pathways that are independent of the permeability transition. TUDCA prevented striatal degeneration and ameliorated locomotor and cognitive deficits in the in vivo 3-nitropropionic acid (3-NP) rat model of HD. Intracellular inclusions were significantly reduced, and the TUDCA-treated mice showed improved locomotor and sensorimotor abilities.

In addition, the antiapoptotic and cytoprotective effects of TUDCA have been tested in models of acute stroke. The possibility that TUDCA exerts an antiapoptotic action by ameliorating mitochondrial function raises the issue whether other neurological disorders, including Friedreich's ataxia, amyotrophic lateral sclerosis, Parkinson's disease, and Alzheimer's disease, can benefit by the administration of TUDCA. This drug is a candidate neuroprotective agent for a variety of chronic neurodegenerative conditions.

ELIGIBILITY:
Inclusion Criteria:

* Caucasian male or female out-patients;
* aged 18 to 75 years inclusive;
* diagnosis of "probable" or "definite" amyotrophic lateral sclerosis according to the El Escorial revised criteria (1);
* first symptoms of ALS by no more than 1.5 years;
* in treatment with steady regimen of riluzole for a minimum of 3 months before study entry, and desiring its continuation;
* FVC ≥ 75% of predicted;
* no conditions known to be contraindications to the use of TUDCA;
* written informed consent.

Exclusion Criteria:

* subjects who underwent tracheostomy;
* subjects who underwent resection of gall bladder;
* subjects with signs of conduction blocks of motor nerves, sensory nerves or both on nerve conduction study;
* subjects with clinical signs of dementia;
* subjects with active peptic ulcer;
* subjects with active malignancy;
* subjects with bulbar onset;
* female subjects who are pregnant or lactating
* subjects who have received an experimental drug or have participated in a clinical trial within 3 months prior to screening
* employees of the investigator or study centre with direct involvement in the proposed study or other studies under the direction of that investigator or study centre.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 34 (Actual)
Dates: Start 2008-06; Primary Completion 2011-07 (Actual); Study Completion 2012-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Alberto Albanese, MD, Principal Investigator — Fondazione IRCCS Istituto neurologico Carlo Besta
Locations (1):
- Fondazione IRCCS Istituto neurologico Carlo Besta, Milan, Milan, Italy

REFERENCES:
- [Background] Brooks BR, Miller RG, Swash M, Munsat TL; World Federation of Neurology Research Group on Motor Neuron Diseases. El Escorial revisited: revised criteria for the diagnosis of amyotrophic lateral sclerosis. Amyotroph Lateral Scler Other Motor Neuron Disord. 2000 Dec;1(5):293-9. doi: 10.1080/146608200300079536. No abstract available. PMID 11464847
- [Background] Cedarbaum JM, Stambler N, Malta E, Fuller C, Hilt D, Thurmond B, Nakanishi A. The ALSFRS-R: a revised ALS functional rating scale that incorporates assessments of respiratory function. BDNF ALS Study Group (Phase III). J Neurol Sci. 1999 Oct 31;169(1-2):13-21. doi: 10.1016/s0022-510x(99)00210-5. PMID 10540002
- [Background] Leigh PN, Swash M, Iwasaki Y, Ludolph A, Meininger V, Miller RG, Mitsumoto H, Shaw P, Tashiro K, Van Den Berg L. Amyotrophic lateral sclerosis: a consensus viewpoint on designing and implementing a clinical trial. Amyotroph Lateral Scler Other Motor Neuron Disord. 2004 Jun;5(2):84-98. doi: 10.1080/14660820410020187. PMID 15204010
- [Background] Keene CD, Rodrigues CM, Eich T, Chhabra MS, Steer CJ, Low WC. Tauroursodeoxycholic acid, a bile acid, is neuroprotective in a transgenic animal model of Huntington's disease. Proc Natl Acad Sci U S A. 2002 Aug 6;99(16):10671-6. doi: 10.1073/pnas.162362299. Epub 2002 Jul 29. PMID 12149470
- [Background] Benz C, Angermuller S, Otto G, Sauer P, Stremmel W, Stiehl A. Effect of tauroursodeoxycholic acid on bile acid-induced apoptosis in primary human hepatocytes. Eur J Clin Invest. 2000 Mar;30(3):203-9. doi: 10.1046/j.1365-2362.2000.00615.x. PMID 10691996
- [Background] Schoemaker MH, Conde de la Rosa L, Buist-Homan M, Vrenken TE, Havinga R, Poelstra K, Haisma HJ, Jansen PL, Moshage H. Tauroursodeoxycholic acid protects rat hepatocytes from bile acid-induced apoptosis via activation of survival pathways. Hepatology. 2004 Jun;39(6):1563-73. doi: 10.1002/hep.20246. PMID 15185297
- [Background] Miller SD, Greene CM, McLean C, Lawless MW, Taggart CC, O'Neill SJ, McElvaney NG. Tauroursodeoxycholic acid inhibits apoptosis induced by Z alpha-1 antitrypsin via inhibition of Bad. Hepatology. 2007 Aug;46(2):496-503. doi: 10.1002/hep.21689. PMID 17559149
- [Background] Rodrigues CM, Sola S, Sharpe JC, Moura JJ, Steer CJ. Tauroursodeoxycholic acid prevents Bax-induced membrane perturbation and cytochrome C release in isolated mitochondria. Biochemistry. 2003 Mar 18;42(10):3070-80. doi: 10.1021/bi026979d. PMID 12627974
- [Background] Ramalho RM, Ribeiro PS, Sola S, Castro RE, Steer CJ, Rodrigues CM. Inhibition of the E2F-1/p53/Bax pathway by tauroursodeoxycholic acid in amyloid beta-peptide-induced apoptosis of PC12 cells. J Neurochem. 2004 Aug;90(3):567-75. doi: 10.1111/j.1471-4159.2004.02517.x. PMID 15255934
- [Background] Rodrigues CM, Sola S, Nan Z, Castro RE, Ribeiro PS, Low WC, Steer CJ. Tauroursodeoxycholic acid reduces apoptosis and protects against neurological injury after acute hemorrhagic stroke in rats. Proc Natl Acad Sci U S A. 2003 May 13;100(10):6087-92. doi: 10.1073/pnas.1031632100. Epub 2003 Apr 29. PMID 12721362
- [Background] Ramalho RM, Borralho PM, Castro RE, Sola S, Steer CJ, Rodrigues CM. Tauroursodeoxycholic acid modulates p53-mediated apoptosis in Alzheimer's disease mutant neuroblastoma cells. J Neurochem. 2006 Sep;98(5):1610-8. doi: 10.1111/j.1471-4159.2006.04007.x. PMID 16923170
- [Background] Ved R, Saha S, Westlund B, Perier C, Burnam L, Sluder A, Hoener M, Rodrigues CM, Alfonso A, Steer C, Liu L, Przedborski S, Wolozin B. Similar patterns of mitochondrial vulnerability and rescue induced by genetic modification of alpha-synuclein, parkin, and DJ-1 in Caenorhabditis elegans. J Biol Chem. 2005 Dec 30;280(52):42655-42668. doi: 10.1074/jbc.M505910200. Epub 2005 Oct 19. PMID 16239214
- [Background] Sola S, Castro RE, Laires PA, Steer CJ, Rodrigues CM. Tauroursodeoxycholic acid prevents amyloid-beta peptide-induced neuronal death via a phosphatidylinositol 3-kinase-dependent signaling pathway. Mol Med. 2003 Sep-Dec;9(9-12):226-34. doi: 10.2119/2003-00042.rodrigues. PMID 15208744
- [Background] Rudolph G, Kloeters-Plachky P, Sauer P, Stiehl A. Intestinal absorption and biliary secretion of ursodeoxycholic acid and its taurine conjugate. Eur J Clin Invest. 2002 Aug;32(8):575-80. doi: 10.1046/j.1365-2362.2002.01030.x. PMID 12190957
- [Background] Keene CD, Rodrigues CM, Eich T, Linehan-Stieers C, Abt A, Kren BT, Steer CJ, Low WC. A bile acid protects against motor and cognitive deficits and reduces striatal degeneration in the 3-nitropropionic acid model of Huntington's disease. Exp Neurol. 2001 Oct;171(2):351-60. doi: 10.1006/exnr.2001.7755. PMID 11573988
- [Background] Castro RE, Sola S, Ramalho RM, Steer CJ, Rodrigues CM. The bile acid tauroursodeoxycholic acid modulates phosphorylation and translocation of bad via phosphatidylinositol 3-kinase in glutamate-induced apoptosis of rat cortical neurons. J Pharmacol Exp Ther. 2004 Nov;311(2):845-52. doi: 10.1124/jpet.104.070532. Epub 2004 Jun 9. PMID 15190125
- [Background] Ince PG, Tomkins J, Slade JY, Thatcher NM, Shaw PJ. Amyotrophic lateral sclerosis associated with genetic abnormalities in the gene encoding Cu/Zn superoxide dismutase: molecular pathology of five new cases, and comparison with previous reports and 73 sporadic cases of ALS. J Neuropathol Exp Neurol. 1998 Oct;57(10):895-904. doi: 10.1097/00005072-199810000-00002. PMID 9786240
- [Background] Chaudhuri KR, Crump S, al-Sarraj S, Anderson V, Cavanagh J, Leigh PN. The validation of El Escorial criteria for the diagnosis of amyotrophic lateral sclerosis: a clinicopathological study. J Neurol Sci. 1995 May;129 Suppl:11-2. doi: 10.1016/0022-510x(95)00050-c. No abstract available. PMID 7595600
- [Background] Turner MR, Bakker M, Sham P, Shaw CE, Leigh PN, Al-Chalabi A. Prognostic modelling of therapeutic interventions in amyotrophic lateral sclerosis. Amyotroph Lateral Scler Other Motor Neuron Disord. 2002 Mar;3(1):15-21. doi: 10.1080/146608202317576499. PMID 12061944
- [Background] Cleveland DW, Rothstein JD. From Charcot to Lou Gehrig: deciphering selective motor neuron death in ALS. Nat Rev Neurosci. 2001 Nov;2(11):806-19. doi: 10.1038/35097565. No abstract available. PMID 11715057
- [Background] Shaw CE, al-Chalabi A, Leigh N. Progress in the pathogenesis of amyotrophic lateral sclerosis. Curr Neurol Neurosci Rep. 2001 Jan;1(1):69-76. doi: 10.1007/s11910-001-0078-7. PMID 11898502
- [Background] Heath PR, Shaw PJ. Update on the glutamatergic neurotransmitter system and the role of excitotoxicity in amyotrophic lateral sclerosis. Muscle Nerve. 2002 Oct;26(4):438-58. doi: 10.1002/mus.10186. PMID 12362409
- [Background] Sathasivam S, Ince PG, Shaw PJ. Apoptosis in amyotrophic lateral sclerosis: a review of the evidence. Neuropathol Appl Neurobiol. 2001 Aug;27(4):257-74. doi: 10.1046/j.0305-1846.2001.00332.x. PMID 11532157
- [Background] Rizzardini M, Lupi M, Bernasconi S, Mangolini A, Cantoni L. Mitochondrial dysfunction and death in motor neurons exposed to the glutathione-depleting agent ethacrynic acid. J Neurol Sci. 2003 Mar 15;207(1-2):51-8. doi: 10.1016/s0022-510x(02)00357-x. PMID 12614931
- [Background] Robertson J, Kriz J, Nguyen MD, Julien JP. Pathways to motor neuron degeneration in transgenic mouse models. Biochimie. 2002 Nov;84(11):1151-60. doi: 10.1016/s0300-9084(02)00025-1. PMID 12595144
- [Background] Rosen DR. Mutations in Cu/Zn superoxide dismutase gene are associated with familial amyotrophic lateral sclerosis. Nature. 1993 Jul 22;364(6435):362. doi: 10.1038/364362c0. No abstract available. PMID 8332197
- [Background] Shaw CE, Enayat ZE, Chioza BA, Al-Chalabi A, Radunovic A, Powell JF, Leigh PN. Mutations in all five exons of SOD-1 may cause ALS. Ann Neurol. 1998 Mar;43(3):390-4. doi: 10.1002/ana.410430319. PMID 9506558
- [Background] Yang Y, Hentati A, Deng HX, Dabbagh O, Sasaki T, Hirano M, Hung WY, Ouahchi K, Yan J, Azim AC, Cole N, Gascon G, Yagmour A, Ben-Hamida M, Pericak-Vance M, Hentati F, Siddique T. The gene encoding alsin, a protein with three guanine-nucleotide exchange factor domains, is mutated in a form of recessive amyotrophic lateral sclerosis. Nat Genet. 2001 Oct;29(2):160-5. doi: 10.1038/ng1001-160. PMID 11586297
- [Background] Puls I, Jonnakuty C, LaMonte BH, Holzbaur EL, Tokito M, Mann E, Floeter MK, Bidus K, Drayna D, Oh SJ, Brown RH Jr, Ludlow CL, Fischbeck KH. Mutant dynactin in motor neuron disease. Nat Genet. 2003 Apr;33(4):455-6. doi: 10.1038/ng1123. Epub 2003 Mar 10. PMID 12627231
- [Background] Al-Chalabi A, Andersen PM, Nilsson P, Chioza B, Andersson JL, Russ C, Shaw CE, Powell JF, Leigh PN. Deletions of the heavy neurofilament subunit tail in amyotrophic lateral sclerosis. Hum Mol Genet. 1999 Feb;8(2):157-64. doi: 10.1093/hmg/8.2.157. PMID 9931323
- [Background] Friedlander RM. Apoptosis and caspases in neurodegenerative diseases. N Engl J Med. 2003 Apr 3;348(14):1365-75. doi: 10.1056/NEJMra022366. No abstract available. PMID 12672865
- [Background] Waldmeier PC. Prospects for antiapoptotic drug therapy of neurodegenerative diseases. Prog Neuropsychopharmacol Biol Psychiatry. 2003 Apr;27(2):303-21. doi: 10.1016/S0278-5846(03)00025-3. PMID 12657369
- [Background] Worms PM. The epidemiology of motor neuron diseases: a review of recent studies. J Neurol Sci. 2001 Oct 15;191(1-2):3-9. doi: 10.1016/s0022-510x(01)00630-x. PMID 11676986
- [Background] Mandrioli J, Faglioni P, Merelli E, Sola P. The epidemiology of ALS in Modena, Italy. Neurology. 2003 Feb 25;60(4):683-9. doi: 10.1212/01.wnl.0000048208.54755.78. PMID 12601112
- [Background] Emery AE, Holloway S. Familial motor neuron diseases. Adv Neurol. 1982;36:139-47. No abstract available. PMID 7180680
- [Background] Bensimon G, Lacomblez L, Meininger V. A controlled trial of riluzole in amyotrophic lateral sclerosis. ALS/Riluzole Study Group. N Engl J Med. 1994 Mar 3;330(9):585-91. doi: 10.1056/NEJM199403033300901. PMID 8302340
- [Background] Lacomblez L, Bensimon G, Leigh PN, Guillet P, Meininger V. Dose-ranging study of riluzole in amyotrophic lateral sclerosis. Amyotrophic Lateral Sclerosis/Riluzole Study Group II. Lancet. 1996 May 25;347(9013):1425-31. doi: 10.1016/s0140-6736(96)91680-3. PMID 8676624
- [Background] Orrell RW, Lane RJ, Ross M. Antioxidant treatment for amyotrophic lateral sclerosis / motor neuron disease. Cochrane Database Syst Rev. 2005 Jan 25;(1):CD002829. doi: 10.1002/14651858.CD002829.pub3. PMID 15674899
- [Background] Moore DH 2nd, Miller RG. Improving efficiency of ALS clinical trials using lead-in designs. Amyotroph Lateral Scler Other Motor Neuron Disord. 2004 Sep;5 Suppl 1:57-60. doi: 10.1080/17434470410019997. PMID 15512875
- [Background] Miller RG, Munsat TL, Swash M, Brooks BR. Consensus guidelines for the design and implementation of clinical trials in ALS. World Federation of Neurology committee on Research. J Neurol Sci. 1999 Oct 31;169(1-2):2-12. doi: 10.1016/s0022-510x(99)00209-9. PMID 10540001
- [Background] Rowland LP, Shneider NA. Amyotrophic lateral sclerosis. N Engl J Med. 2001 May 31;344(22):1688-700. doi: 10.1056/NEJM200105313442207. No abstract available. PMID 11386269
- [Derived] Elia AE, Lalli S, Monsurro MR, Sagnelli A, Taiello AC, Reggiori B, La Bella V, Tedeschi G, Albanese A. Tauroursodeoxycholic acid in the treatment of patients with amyotrophic lateral sclerosis. Eur J Neurol. 2016 Jan;23(1):45-52. doi: 10.1111/ene.12664. Epub 2015 Feb 9. PMID 25664595

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment is started on eightth of october 2009, in medical clinics (Besta Institute in Milan, University II department of Neurology of Naples, University of Palermo department of Neurology).
Pre-assignment Details: 34 patients enrolled, 5 of whom dropped out during the lead in phase.
Groups:
- Placebo: excipient lactose
  Placebo: identical placebo by oral route at the same dosing schedule composed of excipient lactose
Period: Overall Study
Arm/Group | TUDCA | Placebo
Started | 17 | 17
Completed | 15 | 14
Not Completed | 2 | 3

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | TUDCA | Placebo | Total
Number analyzed (Participants) | 17 | 17 | 34
Age, Continuous [Mean (Standard Deviation); unit: years] | 54.0 (12.2) | 58.2 (12.9) | 56.1 (12.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6 | 7 | 13
  Male | 11 | 10 | 21
Region of Enrollment [Number; unit: participants]
  Italy | 17 | 17 | 34

OUTCOME MEASURES:

1. Primary Outcome: The Proportion of Responder Patients in the Two Treatment Groups According the Amyotrophic Lateral Sclerosis Functional Rating Scale (ALSFRS)-R Slope.
Description: Responder patients were defined as those subjects showing an improvement of at least 15% in the ALSFRS-R slope during the treatment period as compared to the lead-in period.
Time Frame: 1 year
Measure: Number; unit: participants
Arm/Group | TUDCA | Placebo
Number analyzed (Participants) | 15 | 14
participants | 13 | 6

2. Secondary Outcome: Forced Vital Capacity (FVC) %
Time Frame: 1 year
Reporting Status: Not Posted

3. Secondary Outcome: SF-36 Quality of Life Rating Scale
Time Frame: 1 year
Reporting Status: Not Posted

4. Secondary Outcome: Time to Tracheostomy From Starting of Study Medication Dosing (if Appropriate)
Time Frame: 1 year
Reporting Status: Not Posted

5. Secondary Outcome: Survival Time From Starting of Study Medication Dosing (if Appropriate)
Time Frame: 1 year
Reporting Status: Not Posted

6. Secondary Outcome: ALSFRS-R at Study End
Time Frame: 1 year
Reporting Status: Not Posted

7. Secondary Outcome: Incidence and Severity of Adverse Events, and Their Relationship to Treatment
Description: laboratory tests, patients' reports and the investigator's judgments
Time Frame: 1 year
Reporting Status: Not Posted

8. Secondary Outcome: Medical Research Council Scores for Right and Left Muscle Groups
Time Frame: 1 year
Reporting Status: Not Posted

ADVERSE EVENTS:
Arm/Group | TUDCA | Placebo
Serious Adverse Events (participants affected / at risk) | 0/15 | 0/14
Other Adverse Events (participants affected / at risk) | 0/15 | 0/14

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No